CLINICAL TRIAL: NCT07300696
Title: Functional Magnetic Resonance Imaging of the Lung to Detect Regional Reversibility and Progression in Interstitial Lung Disease
Brief Title: Functional MRI for Monitoring Progression and Assessing Trends in ILD
Acronym: IMPACT-ILD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: German Center for Lung Research (Other); Thoraxklinik-Heidelberg gGmbH (Other); University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Hans-Ulrich Kauczor, Medical Director of Diagnostic and Interventional Radiology at the Heidelberg University Hospital, University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S-296/2024
Record Dates: First submitted 2025-11-20; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Interstitial Lung Diseases (ILD)
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI Examination Protocol (Experimental)
  Interventions: Diagnostic Test: Lung MRI Protocol with Functional and Contrast-Enhanced Sequences

INTERVENTIONS:
Diagnostic Test: Lung MRI Protocol with Functional and Contrast-Enhanced Sequences — Participants will undergo a lung MRI protocol consisting of structural imaging, non-contrast functional imaging, and contrast-enhanced imaging. Some sequences are custom-developed and performed during free breathing to accommodate patients with respiratory limitations.

SUMMARY:
The main objective of this study is to investigate the utility of functional MRI to differentiate, characterize, and monitor subgroups of ILD. This can be broken down into three specific objectives:

Determine if ILD features observed on high-resolution computed tomography (HRCT), such as ground glass opacities (GGO), are functionally different.

Analyse MRI metrics within each subgroup to determine whether these metrics distinguish different ILDs.

Assess MRI metrics longitudinally to see if these parameters change with disease progression, stability, or reversibility.

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication for a routine HRCT because of either newly diagnosed idiopathic pulmonary fibrosis (IPF) or hypersensitivity pneumonitis (HP) or idiopathic non-specific interstitial pneumonia (iNSIP), suspected diagnosis, or follow-up
* Capacity to consent
* Ability to participate fully in the study (defined by the ability to lie still for the duration of imaging)

Exclusion Criteria:

* Pregnancy and breast feeding
* Persons under the age of 18 and persons not able to give informed consent
* Any medical conditions that could hinder the ability to adhere to the protocol
* Any MRI contraindication, including previous allergic reactions to Gd-based MRI contrast material and renal dysfunction (eGFR < 30 ml min/1,73 m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Identification of ILD Subtypes Using Baseline MRI Metrics | Baseline (first MRI scan)
  Assess whether baseline MRI metrics can accurately differentiate subtypes of interstitial lung disease, using clinician diagnosis (based on multidisciplinary discussion) as the reference standard.

SECONDARY OUTCOMES:
Correlation of Longitudinal MRI Changes with Disease Progression | From enrollment (baseline MRI) through up to 1-year after enrollment; follow-up assessments will only be performed if clinically indicated.
  Evaluate changes in MRI metrics over time and their correlation with ILD progression, using ATS/ERS/JRS/ALAT criteria.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Thoraxklink Heidelberg - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel